CLINICAL TRIAL: NCT00821717
Title: A Randomised, Controlled, Observer-blinded Phase III Clinical Trial to Compare the Effect of Intravenous Ferric Carboxymaltose to Placebo on Exercise Capacity and Cardiac Function in Patients With Chronic Heart Failure and Iron Deficiency
Brief Title: EFfect of Ferric Carboxymaltose on exercIse CApacity and Cardiac Function in Patients With Iron deficiencY and Chronic Heart Failure
Acronym: EFFICACY-HF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Positive FAIR-HF study data are available, this study is identical as EFFICACY-HF. Due to low recruitment in EFFICACY-HF the decision was made to terminate it.
Sponsor: Vifor Pharma (Industry)
Collaborators: Socar Research SA (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FER-CARS-03
Record Dates: First submitted 2009-01-07; First posted 2009-01-13 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Heart Failure; Iron Deficiency; Iron Deficiency Anemia; Anaemia
Keywords: Chronic Heart Failure; Iron deficiency; Iron deficiency anaemia; Anaemia; Heart disease
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency; Anemia; Heart Diseases | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: (Experimental)
  Interventions: Drug: Ferinject ® (Ferric carboxymaltose)
- 2 (Placebo Comparator)
  Interventions: Drug: Normal saline (0.9%)

INTERVENTIONS:
Drug: Ferinject ® (Ferric carboxymaltose) — Ferinject® will be administered in doses of 200 mg (4 mL) weekly up to iron repletion (correction phase of variable duration depending on individual iron deficit). The calculated dose will be rounded to the next 100 mg iron, i.e. the final dose may be 100 mg iron depending on the individual iron deficit.
  After the correction phase, Ferinject® will be given monthly in doses of 200 mg until the 24th week (maintenance phase).
  Arms: 1:
Drug: Normal saline (0.9%) — During the correction phase, patients will receive the number of normal saline injections (4 mL weekly) corresponding to the calculated total iron dose needed according to the individual iron deficit. During the maintenance phase, placebo patients will receive 4 mL normal saline monthly.
  Arms: 2

SUMMARY:
This study is designed to assess, relative to placebo, the effects on the evolution of exercise capacity and symptomatic status of the addition of iron treatment with FCM (ferric carboxymaltose) to the basic regimen of ambulatory patients with stable symptomatic chronic CHF (congestive heart failure) and iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* In New York Heart Association (NYHA) II-III functional class due to stable symptomatic chronic heart failure (CHF)
* Left ventricular ejection fraction (LVEF) 40% or lower for patients in NYHA II and 45% or lower in NYHA III
* Screening haemoglobin (Hb) at least 9.5 g/dL but below or equal to 13.5 g/dL (average of 2 haemoglobin concentrations)
* Screening ferritin below 100 µg/L, or below 300 µg/L when transferrin saturation (TSAT) is below 20%

Exclusion Criteria:

* History of acquired iron overload.
* Known active infection, clinically significant bleeding, active malignancy.
* Chronic liver disease and/or screening alanine transaminase (ALT) or aspartate transaminase (AST)
* Anaemia due to reasons other than iron deficiency
* Immunosuppressive therapy or renal dialysis (current or planned within the next 6 months).
* History of erythropoietin, i.v. or oral iron therapy, and blood transfusion in previous 12 weeks and/or such therapy planned within the next 6 months.
* Unstable angina pectoris as judged by the investigator, clinically significant uncorrected valvular disease or left ventricular outflow obstruction, obstructive cardiomyopathy, poorly controlled fast atrial fibrillation or flutter, poorly controlled symptomatic brady- or tachyarrhythmias.
* Acute myocardial infarction or acute coronary syndrome, transient ischaemic attack or stroke within the last 3 months.
* Coronary-artery bypass graft, percutaneous intervention (e.g. cardiac, cerebrovascular, aortic; diagnostic catheters are allowed) or major surgery, including thoracic and cardiac surgery, within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The distance covered in six-minute walk tests performed at 4, 12 and 24 weeks | 24 weeks
NYHA class assessed at weeks 4, 12 and 24 after the start of study treatment | 24 weeks

SECONDARY OUTCOMES:
Cardiac function assessed by 2D Echo/Doppler cardiography | 24 weeks
Self-reported patient global assessment of treatment | 24 weeks
QOL as assessed by the European Quality of Life - 5 Dimensions and Kansas City Cardi | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Motro, MD, FACC, Study Chair — Sheba Medical Center, Tel-Hashomer 52621, Israel
Locations (41):
- Denmark (8):
  - Research Site, Copenhagen S
  - Research Site, Esbjerg
  - Research Site, Fredericia
  - Research Site, Glostrup Municipality
  - Research Site, Hellerup
  - Research Site, Herning
  - Research Site, Hilleroed
  - Research Site, Svendborg
- France (9):
  - Research Site, Boulogne
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Pontoise
  - Research Site, Rennes
  - Research Site, Saintes
  - Research Site, Strasbourg
- Germany (6):
  - Research Site, Cologne
  - Research Site, Düren
  - Research Site, Frankfurt
  - Research Site, Homburg/Saar
  - Research Site, Mainz
  - Research Site, Würzburg
- Israel (10):
  - Research Site, Afula
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Rehovot
  - Research Site, Safed
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Netherlands (8):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Eindhoven
  - Research Site, Heerenveen
  - Research Site, Leiden
  - Research Site, Nieuwegein
  - Research Site, Tilburg
  - Research Site, Utrecht